CLINICAL TRIAL: NCT07311928
Title: HELIOS: Human Embryo Illumination to Enhance Development
Acronym: HELIOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Samuel Zev Williams, Director of Columbia University Fertility Center; Wendy D. Havens Associate Professor of Women's Health; Chief of the Division of Reproductive Endocrinology and Infertility at Columbia University Irving Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAV9656
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: IVF Outcomes
Keywords: infertility; embryo arrest; recurrent implantation failure; recurrent pregnancy loss; fertility; sperm dna fragmentation
MeSH Terms: conditions — Infertility | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, sibling-embryo-randomized, double-blind controlled trial. All participants will receive the same treatment (IVF/ICSI cycle with PGT-A). Each participant's resultant embryos will be randomized into two groups (one group receiving PBM, the other not).
Who Masked: Participant, Care Provider, Investigator
Masking Description: All embryos will be coded and tracked with blinded identifiers. Embryologists selecting embryos for transfer will be blinded to treatment group. Selection will follow routine morphological and PGT-A criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No photobiomodulation (No Intervention)
- Photobiomodulation (Experimental)
  Interventions: Other: Photobiomodulation

INTERVENTIONS:
Other: Photobiomodulation — Photobiomodulation (PBM), also known as low-level light therapy (LLLT), involves the application of low-intensity red or near-infrared (NIR) light to modulate mitochondrial activity.
  Arms: Photobiomodulation

SUMMARY:
Embryos need a lot of energy to grow, but as women get older, the "power plants" of the cells (called mitochondria) don't work as well. This makes it harder for embryos to develop normally. One possible way to help is with a gentle light treatment called photobiomodulation (PBM). This uses a special type of red light that boosts energy production in cells and helps them stay healthy. This study will test whether adding this light treatment during in vitro fertilization (IVF) can improve embryo growth and pregnancy chances.

DETAILED DESCRIPTION:
Embryo development is highly energy-dependent, and impaired mitochondrial function is a well-established hallmark of reproductive aging. As women age, reactive oxygen species (ROS) accumulate and cause mitochondrial DNA (mtDNA) damage, leading to reduced oxidative phosphorylation, ATP (Adenosine 5'-triphosphate) depletion, and developmental arrest of embryos. Enhancing mitochondrial function represents a promising strategy to improve embryo quality, particularly in women of advanced maternal age.

Photobiomodulation (PBM), also known as low-level light therapy (LLLT), involves the application of low-intensity red or near-infrared (NIR) light to modulate mitochondrial activity. NIR light specifically activates cytochrome c oxidase, leading to increased ATP production, reduced oxidative stress, and improved cellular resilience. Numerous preclinical studies, including isolated mitochondria, cell cultures, and in vivo animal models, have confirmed the safety and efficacy of NIR light in restoring mitochondrial function without inducing DNA damage or chromosomal abnormalities.

The investigators previously conducted IRB-approved laboratory studies using mouse and donated human embryos, demonstrating that brief exposure to PBM improved blastocyst formation without adversely affecting chromosomal status.

The current study builds upon this foundational work to evaluate the clinical impact of PBM during embryo culture in IVF. In a randomized, blinded, sibling-embryo design, the investigators will test whether PBM improves blastocyst formation, embryo quality, and pregnancy outcomes in participants undergoing IVF or ICSI (Intracytoplasmic sperm injection) with PGT-A (preimplantation genetic testing for aneuploidy) using their autologous oocytes.

ELIGIBILITY:
Inclusion Criteria:

* Female age between 18-48 years at time of IVF/ICSI cycle
* Undergoing blastocyst culture and PGT-A
* Using own oocytes
* Have at least two fertilized eggs available for randomization
* Consenting to embryo-level randomization
* Plan to transfer euploid embryo within 6 months

Exclusion Criteria:

* Use of donor eggs
* Known uterine or genetic anomalies
* Refusal of randomization or request for non-standard handling

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of usable blastocysts | Seven days after egg retrieval
  Usable blastocysts are defined as blastocysts that can be biopsied and frozen on Day 5, 6, or 7 of development for PGT-A testing (preimplantation genetic testing for aneuploidy).

SECONDARY OUTCOMES:
Time to 2-cell stage | Up to seven days post egg retrieval
  Time (hours) for embryo to reach the 2-cell stage from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Time to 3-cell stage | Up to seven days post egg retrieval
  Time (hours) for embryo to reach the 3-cell stage from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Time to 6-cell stage | Up to seven days post egg retrieval
  Time (hours) for embryo to reach the 6-cell stage from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Time to 8-cell stage | Up to seven days post egg retrieval
  Time (hours) for embryo to reach the 8-cell stage from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Time to morula | Up to seven days post egg retrieval
  Time (hours) for embryo to reach the morula stage from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Time to start of blastulation | Up to seven days post egg retrieval
  Time (hours) for embryo to start blastulation from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Time to blastocyst | Up to seven days post egg retrieval
  Time (hours) for embryo to reach the blastocyst stage from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Time to hatching blastocyst | Up to seven days post egg retrieval
  Time (hours) for embryo to reach the hatching blastocyst stage from insemination/ICSI as assessed by embryology using Time-lapse imaging.
Number of good quality blastocysts as defined by the Gardner grading system | Up to seven days post egg retrieval
  Final blastocyst quality at the time of cryopreservation (Day 5, 6, or 7) will be assessed using the Gardner grading system, which consists of three parameters: expansion and hatching status (graded 1 - 6), inner cell mass (graded A - D) and trophectoderm (graded A D). A good-quality blastocyst will be defined as a blastocyst of grade 3BB or higher.
Euploidy Rate | Within 30 days post egg retrieval
  The chromosomal ploidy status of cryopreserved blastocysts is assessed as the presence of two copies of each autosome and the expected complement of sex chromosomes. The euploidy rate is defined as the number of cryopreserved blastocysts that have the correct number of chromosomes divided by the total number of cryopreserved blastocysts.
Proportion of Embryo Selected for Transfer | Within 1 year post egg retrieval
  In cases with no stated embryo sex preference, the proportion of cycles in which the embryo selected for transfer is from the PBM-treated group versus the control group will be reported.
Implantation rate | Within 1 year post egg retrieval
  Implantation rate is defined as the number of cycles with positive beta hCG (human chorionic gonadotropin) nine days or more post frozen embryo transfer divided by the total number of frozen embryo transfer cycles.
Clinical pregnancy rate | Within 1 year post egg retrieval
  Clinical pregnancy rate is defined as the number of cycles with the presence of a gestational sac visualized on transvaginal ultrasound divided by the total number of frozen embryo transfer cycles.
Miscarriage rate | Within 1 year of egg retrieval
  Miscarriage rate is defined as number of cycles with clinical pregnancy losses divided by number of cycles that had positive hCGs post frozen embryo transfer.
Live Birth Rate | Up to two years post egg retrieval
  Live birth rate is defined as the number of cycles with a live born infant after 24 weeks gestation divided by the total number of frozen embryo transfer cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Zev Williams, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Fertility Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes